CLINICAL TRIAL: NCT00922207
Title: A Randomized, Open-label Study of the Effect of Peginterferon Alfa-2a (40KD)(PEGASYS) in Combination With Adefovir or Entecavir on HBeAg Seroconversion in Patients With HBeAg Positive Chronic Hepatitis B
Brief Title: A Study of PEGASYS (Peginterferon Alfa-2a (40KD)) in Combination With Adefovir or Entecavir in Patients With HBeAg-Positive Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML21827
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — adefovir; entecavir; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Adefovir; Drug: peginterferon alfa-2a [Pegasys]
- 2 (Experimental)
  Interventions: Drug: Entecavir; Drug: peginterferon alfa-2a [Pegasys]
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: Adefovir — From week -4 to week 2
  Arms: 1
Drug: Entecavir — From week -4 to week 2
  Arms: 2
Drug: Placebo — From week -4 to week 2
  Arms: 3
Drug: peginterferon alfa-2a [Pegasys] — 180 micrograms sc weekly, from week 1-48

SUMMARY:
This 3 arm study will assess the efficacy and safety of PEGASYS alone, or in combination with Adefovir or Entecavir in patients with HBeAg positive chronic hepatitis B. Patients will be randomized to receive 1)PEGASYS 180 micrograms sc weekly for 48 weeks + placebo from weeks -4 to 2;2)PEGASYS 180 micrograms sc weekly for 48 weeks + Adefovir from weeks -4 to 2; or 3)PEGASYS 180 micrograms sc weekly for 48 weeks + Entecavir from weeks -4 to 2. Treatment will be followed by 24 weeks of treatment-free follow-up.The anticipated time on study treatment is 1 year, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-65 years of age;
* HBeAg+ve for >=3 months;
* positive serum HBV DNA within 3 months prior to entry;
* patients with chronic hepatitis B, either naive to HBV treatment, or not responded/relapsed to nucleoside analogues;
* >=3 months treatment-free interval from nucleotide analogues.

Exclusion Criteria:

* evidence of decompensated liver disease;
* history or other evidence of a medical condition associated with chronic liver disease othr than viral hepatitis;
* co-infection with active hepatitis A,C or D, or HIV.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2010-05-07 (Actual); Primary Completion 2014-09-29 (Actual); Study Completion 2014-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Taiwan (9):
  - Changhua Christian Hospital; Internal Medicine, Changhua
  - Kaohsiung Chang Gung Memorial Hospital; Dept of Internal Medicine, Kaohsiung City
  - Kaohsiung Medical Uni Chung-Ho Memorial Hospital; Dept of Internal Medicine, Kaohsiung City
  - Chang Gung Medical Foundation - Keelung; Dept. of Hepato-Gastroenterology, Keelung
  - China Medical University Hospital; Department of Rheumatology, Taichung
  - National Taiwan Uni Hospital; Gastro-Enterology Dept., Taipei
  - Taipei Veterans General Hospital; Gastroenterology Division, Taipei
  - Tri-Service Hospital; Dept. of Internal Medicine, Taipei
  - Chang Gung Medical Foundation - Linkou; Dept. of Hepato-Gastroenterology, Taoyuan District

RESULTS

PARTICIPANT FLOW:
Groups:
- Peg-IFN-Alfa-2a + Adefovir: Participants received adefovir (Hepsera) 10 milligrams (mg) tablet and placebo matched to entecavir tablet, orally once daily for 4 weeks, followed by adefovir 10 mg tablet and placebo matched to entecavir tablet, orally once daily and peginterferon alfa-2a (peg-IFN-alfa-2a; Pegasys) 180 micrograms (µg) subcutaneous (SC) injection once per week, for 2 weeks and then peg-IFN-alfa-2a 180 µg SC injection once per week for 46 weeks.
- Peg-IFN-Alfa-2a + Entecavir: Participants received entecavir (Baraclude) 0.5 mg tablet and placebo matched to adefovir tablet, orally once daily for 4 weeks, followed by entecavir 0.5 mg tablet and placebo matched to adefovir tablet, orally once daily and peg-IFN-alfa-2a 180 µg SC injection once per week, for 2 weeks and then peg-IFN-alfa-2a 180 µg SC injection once per week for 46 weeks.
- Peg-IFN-Alfa-2a + Placebo: Participants received placebo matched to adefovir tablet and placebo matched to entecavir tablet, orally once daily for 4 weeks, followed by placebo matched to adefovir tablet and placebo matched to entecavir tablet, orally once daily and peg-IFN-alfa-2a 180 µg SC injection once per week, for 2 weeks and then peg-IFN-alfa-2a 180 µg SC injection once per week for 46 weeks.
Period: Overall Study
Arm/Group | Peg-IFN-Alfa-2a + Adefovir | Peg-IFN-Alfa-2a + Entecavir | Peg-IFN-Alfa-2a + Placebo
Started | 91 | 95 | 94
Completed | 85 | 88 | 90
Not Completed | 6 | 7 | 4
Not completed — Adverse Event/Intercurrent Illness | 3 | 0 | 0
Not completed — Insufficient Therapeutic Response | 0 | 0 | 1
Not completed — Violation of Selection Criteria at Entry | 0 | 1 | 0
Not completed — Refused Treatment/Did Not Cooperate | 1 | 0 | 0
Not completed — Withdrew Consent | 2 | 5 | 2
Not completed — Abnormality of Laboratory Test | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis population included all randomized participants who received at least one dose of study medication.
Groups:
- Peg-IFN-Alfa-2a + Adefovir: Participants received adefovir 10 mg tablet and placebo matched to entecavir tablet, orally once daily for 4 weeks, followed by adefovir 10 mg tablet and placebo matched to entecavir tablet, orally once daily and peg-IFN-alfa-2a 180 µg SC injection once per week, for 2 weeks and then peg-IFN-alfa-2a 180 µg SC injection once per week for 46 weeks.
- Peg-IFN-Alfa-2a + Entecavir: Participants received entecavir 0.5 mg tablet and placebo matched to adefovir tablet, orally once daily for 4 weeks, followed by entecavir 0.5 mg tablet and placebo matched to adefovir tablet, orally once daily and peg-IFN-alfa-2a 180 µg SC injection once per week, for 2 weeks and then peg-IFN-alfa-2a 180 µg SC injection once per week for 46 weeks.
- Total: Total of all reporting groups
Arm/Group | Peg-IFN-Alfa-2a + Adefovir | Peg-IFN-Alfa-2a + Entecavir | Peg-IFN-Alfa-2a + Placebo | Total
Number analyzed (Participants) | 91 | 95 | 94 | 280
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (9.7) | 37.7 (10.0) | 38.2 (9.7) | 38.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 28 | 81
  Male | 66 | 67 | 66 | 199

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hepatitis B e-Antigen (HBeAg) Seroconversion at 100 Weeks After Start of Treatment
Description: HBeAg seroconversion was defined as the absence of HBeAg (a negative result for HBeAg) and the presence of hepatitis B e-antibody (anti-HBe/HBeAb) (a positive result for anti-HBe).
Time Frame: Week 100
Population: ITT analysis population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peg-IFN-Alfa-2a + Adefovir | Peg-IFN-Alfa-2a + Entecavir | Peg-IFN-Alfa-2a + Placebo
Number analyzed (Participants) | 84 | 88 | 91
percentage of participants | 27.4 [17.8 to 36.9] | 29.5 [20.0 to 39.1] | 36.3 [26.4 to 46.1]
Statistical Analysis 1: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Test type: Superiority or Other; p = 0.6853, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.46 to 1.75]
Statistical Analysis 2: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Test type: Superiority or Other; p = 0.1977, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.35 to 1.26]
Statistical Analysis 3: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Test type: Superiority or Other; p = 0.2916, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.39 to 1.38]

2. Secondary Outcome: Change From Baseline in Hepatitis B Virus Deoxyribonucleic Acid (HBV DNA) Levels at Weeks 4, 8, 16, 28, 40, 52, 64, 76, 88, and 100
Description: HBV DNA (copies per milliliter [copies/mL]) represented the viral load for Hepatitis B Virus (HBV), and was considered an indicator of viral replication.
Time Frame: Baseline, Weeks 4, 8, 16, 28, 40, 52, 64, 76, 88, and 100
Population: ITT analysis population. Here, n = participants who had available assessment at specified time-point.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Peg-IFN-Alfa-2a + Adefovir | Peg-IFN-Alfa-2a + Entecavir | Peg-IFN-Alfa-2a + Placebo
Number analyzed (Participants) | 91 | 95 | 94
copies/mL
  Baseline (n=91,95,94) | 8.65 (1.03) | 8.30 (1.21) | 8.41 (0.96)
  Change at Week 4 (n=90,94,92) | -2.15 (0.94) | -2.76 (0.97) | -0.23 (0.88)
  Change at Week 8 (n=90,94,92) | -1.87 (1.40) | -3.58 (1.12) | -1.32 (1.32)
  Change at Week 16 (n=90,94,92) | -2.14 (1.72) | -3.77 (1.53) | -2.13 (1.93)
  Change at Week 28 (n=90,94,92) | -2.34 (1.90) | -3.07 (1.88) | -2.84 (2.14)
  Change at Week 40 (n=90,94,92) | -2.61 (2.11) | -2.97 (2.11) | -3.27 (2.25)
  Change at Week 52 (n=90,94,92) | -2.75 (2.29) | -2.81 (2.43) | -3.32 (2.48)
  Change at Week 64 (n=90,94,92) | -1.87 (2.26) | -1.37 (2.31) | -2.11 (2.42)
  Change at Week 76 (n=90,94,92) | -1.91 (2.24) | -1.39 (2.46) | -2.20 (2.57)
  Change at Week 88 (n=90,94,92) | -1.78 (2.36) | -1.39 (2.42) | -2.30 (2.34)
  Change at Week 100 (n=90,94,92) | -2.00 (2.35) | -1.78 (2.41) | -2.17 (2.44)
Statistical Analysis 1: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Baseline; Test type: Superiority or Other; p = 0.0353, ANCOVA; Least Squares (LS) Mean Difference = 0.34, 95% CI 2-sided [0.02 to 0.66]
Statistical Analysis 2: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Baseline; Test type: Superiority or Other; p = 0.1114, ANCOVA; LS Mean Difference = 0.23, 95% CI 2-sided [-0.05 to 0.52]
Statistical Analysis 3: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Baseline; Test type: Superiority or Other; p = 0.5150, ANCOVA; LS Mean Difference = -0.10, 95% CI 2-sided [-0.42 to 0.21]
Statistical Analysis 4: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Change at Week 4; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 0.62, 95% CI 2-sided [0.34 to 0.89]
Statistical Analysis 5: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 4; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.92, 95% CI 2-sided [-2.19 to -1.65]
Statistical Analysis 6: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 4; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -2.54, 95% CI 2-sided [-2.81 to -2.27]
Statistical Analysis 7: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Change at Week 8; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.70, 95% CI 2-sided [1.34 to 2.06]
Statistical Analysis 8: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 8; Test type: Superiority or Other; p = 0.0071, ANCOVA; LS Mean Difference = -0.55, 95% CI 2-sided [-0.95 to -0.15]
Statistical Analysis 9: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 8; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -2.26, 95% CI 2-sided [-2.61 to -1.90]
Statistical Analysis 10: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Change at Week 16; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.62, 95% CI 2-sided [1.16 to 2.08]
Statistical Analysis 11: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 16; Test type: Superiority or Other; p = 0.9557, ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.56 to 0.53]
Statistical Analysis 12: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 16; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.65, 95% CI 2-sided [-2.15 to -1.14]
Statistical Analysis 13: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Change at Week 28; Test type: Superiority or Other; p = 0.0094, ANCOVA; LS Mean Difference = 0.73, 95% CI 2-sided [0.18 to 1.27]
Statistical Analysis 14: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 28; Test type: Superiority or Other; p = 0.0943, ANCOVA; LS Mean Difference = 0.51, 95% CI 2-sided [-0.09 to 1.11]
Statistical Analysis 15: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 28; Test type: Superiority or Other; p = 0.4354, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.82 to 0.35]
Statistical Analysis 16: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Change at Week 40; Test type: Superiority or Other; p = 0.2509, ANCOVA; LS Mean Difference = 0.36, 95% CI 2-sided [-0.26 to 0.98]
Statistical Analysis 17: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 40; Test type: Superiority or Other; p = 0.0429, ANCOVA; LS Mean Difference = 0.67, 95% CI 2-sided [0.02 to 1.31]
Statistical Analysis 18: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 40; Test type: Superiority or Other; p = 0.3585, ANCOVA; LS Mean Difference = 0.30, 95% CI 2-sided [-0.34 to 0.93]
Statistical Analysis 19: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Change at Week 52; Test type: Superiority or Other; p = 0.9014, ANCOVA; LS Mean Difference = 0.04, 95% CI 2-sided [-0.65 to 0.74]
Statistical Analysis 20: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 52; Test type: Superiority or Other; p = 0.1122, ANCOVA; LS Mean Difference = 0.57, 95% CI 2-sided [-0.13 to 1.28]
Statistical Analysis 21: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 52; Test type: Superiority or Other; p = 0.1602, ANCOVA; LS Mean Difference = 0.51, 95% CI 2-sided [-0.20 to 1.23]
Statistical Analysis 22: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Change at Week 64; Test type: Superiority or Other; p = 0.1599, ANCOVA; LS Mean Difference = -0.49, 95% CI 2-sided [-1.17 to 0.19]
Statistical Analysis 23: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 64; Test type: Superiority or Other; p = 0.5045, ANCOVA; LS Mean Difference = 0.23, 95% CI 2-sided [-0.45 to 0.92]
Statistical Analysis 24: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 64; Test type: Superiority or Other; p = 0.0412, ANCOVA; LS Mean Difference = 0.72, 95% CI 2-sided [0.03 to 1.41]
Statistical Analysis 25: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Change at Week 76; Test type: Superiority or Other; p = 0.1347, ANCOVA; LS Mean Difference = -0.54, 95% CI 2-sided [-1.24 to 0.17]
Statistical Analysis 26: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 76; Test type: Superiority or Other; p = 0.4027, ANCOVA; LS Mean Difference = 0.30, 95% CI 2-sided [-0.41 to 1.01]
Statistical Analysis 27: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 76; Test type: Superiority or Other; p = 0.0311, ANCOVA; LS Mean Difference = 0.81, 95% CI 2-sided [0.07 to 1.55]
Statistical Analysis 28: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Change at Week 88; Test type: Superiority or Other; p = 0.3183, ANCOVA; LS Mean Difference = -0.36, 95% CI 2-sided [-1.07 to 0.35]
Statistical Analysis 29: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 88; Test type: Superiority or Other; p = 0.1371, ANCOVA; LS Mean Difference = 0.52, 95% CI 2-sided [-0.17 to 1.22]
Statistical Analysis 30: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 88; Test type: Superiority or Other; p = 0.0113, ANCOVA; LS Mean Difference = 0.90, 95% CI 2-sided [0.21 to 1.60]
Statistical Analysis 31: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 100; Test type: Superiority or Other; p = 0.5608, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.92 to 0.50]
Statistical Analysis 32: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 100; Test type: Superiority or Other; p = 0.6323, ANCOVA; LS Mean Difference = 0.17, 95% CI 2-sided [-0.53 to 0.88]
Statistical Analysis 33: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 100; Test type: Superiority or Other; p = 0.2752, ANCOVA; LS Mean Difference = 0.40, 95% CI 2-sided [-0.32 to 1.11]

3. Secondary Outcome: Percentage of Participants Who Were HBeAg Negative
Time Frame: Baseline, Weeks 4, 8, 16, 28, 40, 52, 64, 76, 88, and 100
Population: ITT analysis population. Here, n = participants who had available assessment at specified time-point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peg-IFN-Alfa-2a + Adefovir | Peg-IFN-Alfa-2a + Entecavir | Peg-IFN-Alfa-2a + Placebo
Number analyzed (Participants) | 91 | 95 | 94
percentage of participants
  Baseline (n=91,95,94) | 3.3 [0.0 to 7.0] | 2.1 [0.0 to 5.0] | 0.0 [NA to NA] — The 95 percent (%) confidence interval (CV) could not be calculated as no participant had response at this time-point.
  Week 4 (n=90,94,92) | 5.6 [0.8 to 10.3] | 4.3 [0.2 to 8.3] | 1.1 [0.0 to 3.2]
  Week 8 (n=90,94,92) | 6.7 [1.5 to 11.8] | 6.4 [1.4 to 11.3] | 4.3 [0.2 to 8.5]
  Week 16 (n=90,94,92) | 6.7 [1.5 to 11.8] | 8.5 [2.9 to 14.2] | 10.9 [4.5 to 17.2]
  Week 28 (n=90,94,92) | 11.1 [4.6 to 17.6] | 10.6 [4.4 to 16.9] | 16.3 [8.8 to 23.9]
  Week 40 (n=90,94,92) | 18.9 [10.8 to 27.0] | 18.1 [10.3 to 25.9] | 22.8 [14.2 to 31.4]
  Week 52 (n=90,94,92) | 22.2 [13.6 to 30.8] | 22.3 [13.9 to 30.8] | 29.3 [20.0 to 38.7]
  Week 64 (n=90,92,92) | 24.4 [15.6 to 33.3] | 25.0 [16.2 to 33.8] | 31.5 [22.0 to 41.0]
  Week 76 (n=88,88,92) | 25.0 [16.0 to 34.0] | 28.4 [19.0 to 37.8] | 37.0 [27.1 to 46.8]
  Week 88 (n=86,87,90) | 27.9 [18.4 to 37.4] | 27.6 [18.2 to 37.0] | 34.4 [24.6 to 44.3]
  Week 100 (n=84,87,91) | 28.6 [18.9 to 38.2] | 32.2 [22.4 to 42.0] | 37.4 [27.4 to 47.3]
Statistical Analysis 1: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Baseline; Test type: Superiority or Other; p = 0.6107, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.59, 95% CI 2-sided [0.26 to 9.71]
Statistical Analysis 2: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Baseline; Test type: Superiority or Other; p = 0.0788, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Baseline; Test type: Superiority or Other; p = 0.1761, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 4; Test type: Superiority or Other; p = 0.7044, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.34 to 5.09]
Statistical Analysis 5: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 4; Test type: Superiority or Other; p = 0.0927, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 5.35, 95% CI 2-sided [0.61 to 46.76]
Statistical Analysis 6: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 4; Test type: Superiority or Other; p = 0.1858, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.04, 95% CI 2-sided [0.44 to 36.89]
Statistical Analysis 7: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 8; Test type: Superiority or Other; p = 0.9385, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.33 to 3.38]
Statistical Analysis 8: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 8; Test type: Superiority or Other; p = 0.5068, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.43 to 5.77]
Statistical Analysis 9: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 8; Test type: Superiority or Other; p = 0.5544, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.41 to 5.50]
Statistical Analysis 10: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 16; Test type: Superiority or Other; p = 0.6510, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.26 to 2.31]
Statistical Analysis 11: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 16; Test type: Superiority or Other; p = 0.3192, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.20 to 1.69]
Statistical Analysis 12: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 16; Test type: Superiority or Other; p = 0.5818, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.29 to 2.03]
Statistical Analysis 13: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 28; Test type: Superiority or Other; p = 0.8796, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.41 to 2.66]
Statistical Analysis 14: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 28; Test type: Superiority or Other; p = 0.3050, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.27 to 1.52]
Statistical Analysis 15: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 28; Test type: Superiority or Other; p = 0.2414, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.26 to 1.44]
Statistical Analysis 16: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 40; Test type: Superiority or Other; p = 0.8502, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.50 to 2.22]
Statistical Analysis 17: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 40; Test type: Superiority or Other; p = 0.5000, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.38 to 1.61]
Statistical Analysis 18: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 40; Test type: Superiority or Other; p = 0.3882, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.36 to 1.53]
Statistical Analysis 19: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 52; Test type: Superiority or Other; p = 0.9584, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.50 to 1.99]
Statistical Analysis 20: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 52; Test type: Superiority or Other; p = 0.2576, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.35 to 1.34]
Statistical Analysis 21: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 52; Test type: Superiority or Other; p = 0.2362, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.36 to 1.34]
Statistical Analysis 22: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 64; Test type: Superiority or Other; p = 0.9861, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.49 to 1.90]
Statistical Analysis 23: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 64; Test type: Superiority or Other; p = 0.2919, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.37 to 1.35]
Statistical Analysis 24: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 64; Test type: Superiority or Other; p = 0.2674, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.38 to 1.38]
Statistical Analysis 25: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 76; Test type: Superiority or Other; p = 0.6148, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.43 to 1.64]
Statistical Analysis 26: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 76; Test type: Superiority or Other; p = 0.0904, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.57, 95% CI 2-sided [0.30 to 1.08]
Statistical Analysis 27: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 76; Test type: Superiority or Other; p = 0.2073, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.36 to 1.27]
Statistical Analysis 28: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 88; Test type: Superiority or Other; p = 0.9980, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.52 to 1.98]
Statistical Analysis 29: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 88; Test type: Superiority or Other; p = 0.3489, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.39 to 1.40]
Statistical Analysis 30: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 88; Test type: Superiority or Other; p = 0.2847, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.38 to 1.38]
Statistical Analysis 31: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 100; Test type: Superiority or Other; p = 0.5596, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.44 to 1.62]
Statistical Analysis 32: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 100; Test type: Superiority or Other; p = 0.2112, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.36 to 1.27]
Statistical Analysis 33: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 100; Test type: Superiority or Other; p = 0.4066, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.43 to 1.48]

4. Secondary Outcome: Percentage of Participant Who Were Both Hepatitis B Surface Antigen (HBsAg) Negative and Hepatitis B Surface Antibody (Anti-HBs/HBsAb) Positive
Time Frame: Baseline, Weeks 4, 8, 16, 28, 40, 52, 64, 76, 88, and 100
Population: ITT analysis population. Here, n = participants who had available assessment at specified time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Peg-IFN-Alfa-2a + Adefovir | Peg-IFN-Alfa-2a + Entecavir | Peg-IFN-Alfa-2a + Placebo
Number analyzed (Participants) | 91 | 95 | 94
percentage of participants
  Baseline (n=91,95,94) | 0.0 | 0.0 | 0.0
  Week 4 (n=90,94,92) | 0.0 | 0.0 | 0.0
  Week 8 (n=90,94,92) | 0.0 | 0.0 | 0.0
  Week 16 (n=90,94,92) | 0.0 | 0.0 | 0.0
  Week 28 (n=90,94,92) | 0.0 | 0.0 | 0.0
  Week 40 (n=90,94,92) | 0.0 | 0.0 | 0.0
  Week 52 (n=90,94,92) | 0.0 | 0.0 | 0.0
  Week 64 (n=90,92,92) | 0.0 | 0.0 | 0.0
  Week 76 (n=88,88,92) | 0.0 | 0.0 | 0.0
  Week 88 (n=86,87,90) | 1.2 | 0.0 | 3.4
  Week 100 (n=84,87,91) | 0.0 | 0.0 | 0.0

5. Secondary Outcome: Percentage of Participant With Normal Alanine Aminotransferase (ALT) Levels
Description: The normal range for ALT is 10 to 40 international units per liter (IU/L).
Time Frame: Baseline, Weeks 6, 12, 16, 22, 28, 34, 40, 46, 52, 64, 76, 88, and 100
Population: ITT analysis population. Here, n = participants who had available assessment at specified time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Peg-IFN-Alfa-2a + Adefovir | Peg-IFN-Alfa-2a + Entecavir | Peg-IFN-Alfa-2a + Placebo
Number analyzed (Participants) | 91 | 95 | 94
percentage of participants
  Baseline (n=91,95,94) | 4.4 | 3.2 | 2.1
  Week 6 (n=90,93,92) | 4.4 | 5.4 | 6.5
  Week 12 (n=90,93,92) | 15.6 | 17.2 | 13.0
  Week 16 (n=90,93,92) | 21.1 | 24.7 | 20.7
  Week 22 (n=90,93,92) | 25.6 | 34.4 | 22.8
  Week 28 (n=90,93,92) | 26.7 | 30.1 | 23.9
  Week 34 (n=90,93,92) | 26.7 | 34.4 | 32.6
  Week 40 (n=90,93,92) | 30.0 | 39.8 | 32.6
  Week 46 (n=90,93,92) | 30.0 | 41.9 | 33.7
  Week 52 (n=90,93,92) | 33.3 | 34.4 | 32.6
  Week 64 (n=90,92,92) | 32.2 | 37.0 | 42.4
  Week 76 (n=89,89,92) | 43.8 | 38.2 | 46.7
  Week 88 (n=86,88,91) | 32.6 | 33.0 | 48.4
  Week 100 (n=84,88,91) | 36.9 | 40.9 | 49.5
Statistical Analysis 1: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Baseline; Test type: Superiority or Other; p = 0.6921, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.41
Statistical Analysis 2: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Baseline; Test type: Superiority or Other; p = 0.3939, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.11
Statistical Analysis 3: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Baseline; Test type: Superiority or Other; p = 0.6818, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.50
Statistical Analysis 4: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 6; Test type: Superiority or Other; p = 0.7582, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.82
Statistical Analysis 5: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 6; Test type: Superiority or Other; p = 0.5381, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.67
Statistical Analysis 6: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 6; Test type: Superiority or Other; p = 0.7747, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.81
Statistical Analysis 7: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 12; Test type: Superiority or Other; p = 0.8034, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.89
Statistical Analysis 8: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 12; Test type: Superiority or Other; p = 0.6306, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.23
Statistical Analysis 9: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 12; Test type: Superiority or Other; p = 0.4574, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.39
Statistical Analysis 10: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 16; Test type: Superiority or Other; p = 0.5824, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.81
Statistical Analysis 11: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 16; Test type: Superiority or Other; p = 0.9321, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.03
Statistical Analysis 12: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 16; Test type: Superiority or Other; p = 0.5263, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.26
Statistical Analysis 13: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 22; Test type: Superiority or Other; p = 0.2025, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.65
Statistical Analysis 14: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 22; Test type: Superiority or Other; p = 0.6702, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.16
Statistical Analysis 15: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 22; Test type: Superiority or Other; p = 0.0818, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.77
Statistical Analysis 16: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 28; Test type: Superiority or Other; p = 0.6214, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.84
Statistical Analysis 17: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 28; Test type: Superiority or Other; p = 0.6774, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.16
Statistical Analysis 18: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 28; Test type: Superiority or Other; p = 0.3154, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.37
Statistical Analysis 19: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 34; Test type: Superiority or Other; p = 0.2709, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.69
Statistical Analysis 20: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 34; Test type: Superiority or Other; p = 0.3804, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.75
Statistical Analysis 21: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 34; Test type: Superiority or Other; p = 0.7645, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.08
Statistical Analysis 22: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 40; Test type: Superiority or Other; p = 0.1820, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.65
Statistical Analysis 23: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 40; Test type: Superiority or Other; p = 0.7167, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.89
Statistical Analysis 24: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 40; Test type: Superiority or Other; p = 0.3104, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.37
Statistical Analysis 25: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 46; Test type: Superiority or Other; p = 0.0910, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.59
Statistical Analysis 26: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 46; Test type: Superiority or Other; p = 0.6094, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.84
Statistical Analysis 27: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 46; Test type: Superiority or Other; p = 0.2166, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.42
Statistical Analysis 28: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 52; Test type: Superiority or Other; p = 0.9010, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.95
Statistical Analysis 29: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 52; Test type: Superiority or Other; p = 0.9060, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.03
Statistical Analysis 30: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 52; Test type: Superiority or Other; p = 0.7268, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.08
Statistical Analysis 31: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 64; Test type: Superiority or Other; p = 0.5372, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.81
Statistical Analysis 32: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 64; Test type: Superiority or Other; p = 0.1588, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.65
Statistical Analysis 33: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 64; Test type: Superiority or Other; p = 0.4268, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.80
Statistical Analysis 34: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 76; Test type: Superiority or Other; p = 0.4389, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.26
Statistical Analysis 35: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 76; Test type: Superiority or Other; p = 0.6708, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.89
Statistical Analysis 36: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 76; Test type: Superiority or Other; p = 0.2145, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.70
Statistical Analysis 37: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 88; Test type: Superiority or Other; p = 0.8608, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.98
Statistical Analysis 38: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 88; Test type: Superiority or Other; p = 0.0283, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.52
Statistical Analysis 39: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 88; Test type: Superiority or Other; p = 0.0369, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.53
Statistical Analysis 40: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Week 100; Test type: Superiority or Other; p = 0.4606, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.84
Statistical Analysis 41: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Week 100; Test type: Superiority or Other; p = 0.0832, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.60
Statistical Analysis 42: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Week 100; Test type: Superiority or Other; p = 0.2655, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.71

6. Secondary Outcome: Change From Baseline in HBsAg Levels at Weeks 4, 8, 16, 28, 40, 52, 64, 76, 88, and 100
Time Frame: Baseline, Weeks 4, 8, 16, 28, 40, 52, 64, 76, 88, and 100
Population: ITT analysis population. Here, n = participants who had available assessment at specified time-point.
Measure: Mean (Standard Deviation); unit: International Units/milliliter (IU/mL)
Arm/Group | Peg-IFN-Alfa-2a + Adefovir | Peg-IFN-Alfa-2a + Entecavir | Peg-IFN-Alfa-2a + Placebo
Number analyzed (Participants) | 91 | 95 | 94
International Units/milliliter (IU/mL)
  Baseline (n=91,95,94) | 3.97 (0.72) | 3.76 (0.83) | 3.84 (0.71)
  Change at Week 4 (n=90,94,92) | -0.26 (0.48) | -0.18 (0.44) | -0.02 (0.33)
  Change at Week 8 (n=90,94,92) | -0.33 (0.78) | -0.31 (0.58) | -0.25 (0.56)
  Change at Week 16 (n=90,94,92) | -0.40 (0.78) | -0.49 (0.74) | -0.48 (0.83)
  Change at Week 28 (n=90,94,92) | -0.61 (0.96) | -0.68 (0.98) | -0.70 (1.08)
  Change at Week 40 (n=90,94,92) | -0.71 (1.09) | -0.67 (1.04) | -0.82 (1.27)
  Change at Week 52 (n=90,94,92) | -0.78 (1.27) | -0.69 (1.11) | -0.88 (1.41)
  Change at Week 64 (n=90,94,92) | -0.67 (1.18) | -0.54 (1.07) | -0.67 (1.21)
  Change at Week 76 (n=90,94,92) | -0.58 (0.95) | -0.45 (1.01) | -0.53 (1.19)
  Change at Week 88 (n=90,94,92) | -0.50 (1.11) | -0.44 (0.90) | -0.62 (1.20)
  Change at Week 100 (n=90,94,92) | -0.41 (0.75) | -0.60 (1.15) | -0.56 (1.10)
Statistical Analysis 1: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Baseline; Test type: Superiority or Other; p = 0.0649, ANCOVA; LS Mean Difference = 0.21, 95% CI 2-sided [-0.01 to 0.43]
Statistical Analysis 2: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Baseline; Test type: Superiority or Other; p = 0.1867, ANCOVA; LS Mean Difference = 0.13, 95% CI 2-sided [-0.06 to 0.33]
Statistical Analysis 3: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Baseline; Test type: Superiority or Other; p = 0.5003, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.30 to 0.15]
Statistical Analysis 4: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Change at Week 4; Test type: Superiority or Other; p = 0.2259, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.22 to 0.05]
Statistical Analysis 5: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 4; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.36 to -0.11]
Statistical Analysis 6: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 4; Test type: Superiority or Other; p = 0.0085, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.27 to -0.04]
Statistical Analysis 7: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Change at Week 8; Test type: Superiority or Other; p = 0.8160, ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.22 to 0.18]
Statistical Analysis 8: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 8; Test type: Superiority or Other; p = 0.4393, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.27 to 0.12]
Statistical Analysis 9: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 8; Test type: Superiority or Other; p = 0.4890, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.22 to 0.11]
Statistical Analysis 10: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Change at Week 16; Test type: Superiority or Other; p = 0.4656, ANCOVA; LS Mean Difference = 0.08, 95% CI 2-sided [-0.14 to 0.30]
Statistical Analysis 11: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 16; Test type: Superiority or Other; p = 0.5016, ANCOVA; LS Mean Difference = 0.08, 95% CI 2-sided [-0.15 to 0.31]
Statistical Analysis 12: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 16; Test type: Superiority or Other; p = 0.9582, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.23 to 0.22]
Statistical Analysis 13: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Change at Week 28; Test type: Superiority or Other; p = 0.6214, ANCOVA; LS Mean Difference = 0.07, 95% CI 2-sided [-0.21 to 0.36]
Statistical Analysis 14: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 28; Test type: Superiority or Other; p = 0.5493, ANCOVA; LS Mean Difference = 0.09, 95% CI 2-sided [-0.21 to 0.39]
Statistical Analysis 15: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 28; Test type: Superiority or Other; p = 0.8881, ANCOVA; LS Mean Difference = 0.02, 95% CI 2-sided [-0.28 to 0.32]
Statistical Analysis 16: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Change at Week 40; Test type: Superiority or Other; p = 0.7912, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.36 to 0.27]
Statistical Analysis 17: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 40; Test type: Superiority or Other; p = 0.5427, ANCOVA; LS Mean Difference = 0.11, 95% CI 2-sided [-0.24 to 0.46]
Statistical Analysis 18: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 40; Test type: Superiority or Other; p = 0.3788, ANCOVA; LS Mean Difference = 0.15, 95% CI 2-sided [-0.19 to 0.49]
Statistical Analysis 19: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Change at Week 52; Test type: Superiority or Other; p = 0.6172, ANCOVA; LS Mean Difference = -0.09, 95% CI 2-sided [-0.44 to 0.26]
Statistical Analysis 20: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 52; Test type: Superiority or Other; p = 0.6002, ANCOVA; LS Mean Difference = 0.11, 95% CI 2-sided [-0.29 to 0.50]
Statistical Analysis 21: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 52; Test type: Superiority or Other; p = 0.3101, ANCOVA; LS Mean Difference = 0.19, 95% CI 2-sided [-0.18 to 0.56]
Statistical Analysis 22: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Change at Week 64; Test type: Superiority or Other; p = 0.4256, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.47 to 0.20]
Statistical Analysis 23: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 64; Test type: Superiority or Other; p = 0.9762, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.35 to 0.36]
Statistical Analysis 24: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 64; Test type: Superiority or Other; p = 0.4504, ANCOVA; LS Mean Difference = 0.13, 95% CI 2-sided [-0.21 to 0.47]
Statistical Analysis 25: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Change at Week 76; Test type: Superiority or Other; p = 0.4076, ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-0.42 to 0.17]
Statistical Analysis 26: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 76; Test type: Superiority or Other; p = 0.7591, ANCOVA; LS Mean Difference = -0.05, 95% CI 2-sided [-0.37 to 0.27]
Statistical Analysis 27: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 76; Test type: Superiority or Other; p = 0.6449, ANCOVA; LS Mean Difference = 0.08, 95% CI 2-sided [-0.25 to 0.40]
Statistical Analysis 28: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Change at Week 88; Test type: Superiority or Other; p = 0.7108, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.36 to 0.25]
Statistical Analysis 29: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 88; Test type: Superiority or Other; p = 0.4725, ANCOVA; LS Mean Difference = 0.12, 95% CI 2-sided [-0.22 to 0.47]
Statistical Analysis 30: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 88; Test type: Superiority or Other; p = 0.2439, ANCOVA; LS Mean Difference = 0.19, 95% CI 2-sided [-0.13 to 0.50]
Statistical Analysis 31: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Entecavir; Change at Week 100; Test type: Superiority or Other; p = 0.1862, ANCOVA; LS Mean Difference = 0.20, 95% CI 2-sided [-0.10 to 0.50]
Statistical Analysis 32: Comparison: Peg-IFN-Alfa-2a + Adefovir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 100; Test type: Superiority or Other; p = 0.3057, ANCOVA; LS Mean Difference = 0.15, 95% CI 2-sided [-0.14 to 0.43]
Statistical Analysis 33: Comparison: Peg-IFN-Alfa-2a + Entecavir vs Peg-IFN-Alfa-2a + Placebo; Change at Week 100; Test type: Superiority or Other; p = 0.8002, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.38 to 0.29]

7. Secondary Outcome: Percentage of Participants With Combined Response
Description: Combined response was defined as having negative HBeAg, HBV DNA less than (<) 100,000 copies/mL, and normal ALT level (10-40 IU/L).
Time Frame: Baseline, Weeks 4, 8, 16, 28, 40, 52, 64, 76, 88, and 100
Population: ITT analysis population. Here, n = participants who had available assessment at specified time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Peg-IFN-Alfa-2a + Adefovir | Peg-IFN-Alfa-2a + Entecavir | Peg-IFN-Alfa-2a + Placebo
Number analyzed (Participants) | 91 | 95 | 94
percentage of participants
  Baseline (n=91,95,94) | 0.0 | 0.0 | 0.0
  Week 16 (n=90,93,92) | 0.0 | 0.0 | 0.0
  Week 28 (n=90,93,92) | 0.0 | 1.1 | 0.0
  Week 40 (n=90,93,92) | 0.0 | 0.0 | 0.0
  Week 52 (n=90,93,92) | 0.0 | 0.0 | 0.0
  Week 64 (n=90,92,92) | 2.2 | 0.0 | 0.0
  Week 76 (n=88,89,92) | 3.4 | 0.0 | 0.0
  Week 88 (n=86,88,91) | 3.5 | 0.0 | 0.0
  Week 100 (n=84,88,91) | 2.4 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 100
Description: Safety analysis population included participants who received at least one dose of study medication and had at least one post-baseline safety assessment.
Arm/Group | Peg-IFN-Alfa-2a + Adefovir | Peg-IFN-Alfa-2a + Entecavir | Peg-IFN-Alfa-2a + Placebo
Serious Adverse Events (participants affected / at risk) | 7/91 | 12/94 | 7/93
Other Adverse Events (participants affected / at risk) | 85/91 | 83/94 | 89/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peg-IFN-Alfa-2a + Adefovir (N=91) | Peg-IFN-Alfa-2a + Entecavir (N=94) | Peg-IFN-Alfa-2a + Placebo (N=93)
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 0
Hepatitis B (Infections and infestations) | 2 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 4 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Calculus urethral (Renal and urinary disorders) | 1 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper gastrointestinal heamorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peg-IFN-Alfa-2a + Adefovir (N=91) | Peg-IFN-Alfa-2a + Entecavir (N=94) | Peg-IFN-Alfa-2a + Placebo (N=93)
Chills (General disorders) | 6 | 0 | 4
Fatigue (General disorders) | 13 | 12 | 15
Influenza like illnes (General disorders) | 3 | 5 | 3
Injection site pain (General disorders) | 4 | 5 | 4
Malaise (General disorders) | 5 | 3 | 5
Pyrexia (General disorders) | 20 | 19 | 21
Hepatic steatosis (Hepatobiliary disorders) | 5 | 2 | 1
Influenza (Infections and infestations) | 4 | 8 | 2
Nasopharyngitis (Infections and infestations) | 8 | 7 | 10
Upper respiratory tract infection (Infections and infestations) | 6 | 11 | 14
Alanine aminotransferase increased (Investigations) | 14 | 17 | 18
Weight decreased (Investigations) | 5 | 9 | 3
Decreased appetite (Metabolism and nutrition disorders) | 8 | 7 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 6 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 13 | 18
Dizziness (Nervous system disorders) | 8 | 14 | 8
Headache (Nervous system disorders) | 21 | 17 | 20
Insomnia (Psychiatric disorders) | 6 | 4 | 11
Neutropenia (Blood and lymphatic system disorders) | 6 | 8 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3 | 6
Abdominal distension (Gastrointestinal disorders) | 7 | 9 | 4
Abdominal pain (Gastrointestinal disorders) | 5 | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 6 | 5 | 6
Diarrhoea (Gastrointestinal disorders) | 14 | 9 | 13
Gingival bleeding (Gastrointestinal disorders) | 3 | 0 | 8
Mouth ulceration (Gastrointestinal disorders) | 4 | 6 | 3
Nausea (Gastrointestinal disorders) | 7 | 10 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 23 | 27 | 25
Eczema (Skin and subcutaneous tissue disorders) | 7 | 1 | 5
Pruritis (Skin and subcutaneous tissue disorders) | 11 | 14 | 15
Rash (Skin and subcutaneous tissue disorders) | 10 | 10 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.